CLINICAL TRIAL: NCT00535496
Title: Comparison of the T4/T1 Ratio Measured by Means of the TOF Watch® SX With the Reappearance of T4 Measured by Means of a Peripheral Nerve Stimulator in Adult Subjects Receiving 4.0 mg.Kg-1 Sugammadex at 15 Minutes After Rocuronium
Brief Title: Relation Between TOF-Watch® SX and a Peripheral Nerve Stimulator After 4.0 mg.Kg-1 Sugammadex (P05698)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05698; 19.4.313
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Results first posted 2013-09-02 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-02

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): sugammadex 1.0 mg/kg, TOF-Watch® SX (dominant forearm) and PNS (non-dominant forearm)
  Interventions: Drug: sugammadex
- 2 (Experimental): sugammadex 1.0 mg/kg, TOF-Watch® SX (non-dominant forearm) and PNS (dominant forearm)
  Interventions: Drug: sugammadex
- 3 (Experimental): sugammadex 4.0 mg/kg, TOF-Watch® SX (dominant forearm) and PNS (non-dominant forearm)
  Interventions: Drug: sugammadex
- 4 (Experimental): sugammadex 4.0 mg/kg, TOF-Watch® SX (non-dominant forearm) and PNS (dominant forearm)
  Interventions: Drug: sugammadex

INTERVENTIONS:
Drug: sugammadex — Participants will receive an intubating dose of 0.6 mg/kg rocuronium, followed by one or more maintenance doses of 0.15 mg/kg rocuronium, if necessary. Fifteen minutes after the last dose of rocuronium, 1.0 or 4.0 mg/kg sugammadex will be randomly administered by intravenous (IV) bolus dose based on actual body weight.
  Other Names: Org 25969; Bridion®; MK-8616; SCH 900616

SUMMARY:
The objective of the trial is to determine the relationship within a participant between the time to manual detection of the reappearance of the fourth twitch (T4) measured using a peripheral nerve stimulator (PNS) and the time to recovery of the fourth twitch/first twitch (T4/T1) ratio to 0.9 measured using a Train Of Four (TOF)-Watch® SX, of 4.0 mg/kg sugammadex administered at 15 minutes after either a bolus dose of 0.6 mg/kg rocuronium or the last maintenance dose of 0.15 mg/kg rocuronium.

DETAILED DESCRIPTION:
The TOF-Watch® SX has been used for neuromuscular monitoring in all

clinical trials with sugammadex. In clinical practice however, a PNS is commonly

used in many hospitals worldwide. A disadvantage of a PNS is that it is not objective monitoring like the TOF-Watch® SX, and it can detect only the number of twitches. In this trial, the relationship between the time to reappearance of T4 using PNS (i.e. Ministim® model MS-IV) and the time to recovery of the T4/T1 ratio to 0.9 using the TOF-Watch® SX was determined after a dose of 4.0 mg/kg sugammadex was administered 15 minutes after the last dose of rocuronium. Determining this relationship will enable the provision of advice on when it is safe to extubate participants after administration of 4.0 mg/kg sugammadex for reversing neuromuscular block while using a PNS. The time to reappearance of T4 was assessed by a blinded PNS-assessor. This assessor was blinded for the dose of sugammadex used and for the TOF results measured with the TOF-Watch® SX.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class 1 or 2 or 3
* between the ages of 18 to 64 years, inclusive
* scheduled for a surgical procedure under general anesthesia requiring

neuromuscular relaxation with the use of rocuronium

* scheduled for a surgical procedure in supine position
* have given written informed consent

Exclusion Criteria:

* participants with a difficult intubation because of expected anatomical

malformations

* known or suspected to have neuromuscular disorders impairing

neuromuscular blockade and/or significant hepatic and/or renal

dysfunction

* medical or physical condition that is expected to interfere

with the proper conduct of simultaneous neuromuscular monitoring on

both arms

* known or suspected to have a (family) history of malignant

hyperthermia

* known or suspected to have arthritis or another disease that will

cause the thumb not to move freely

* known or suspected to have an allergy to narcotics, muscle

relaxants or other medication used during general anesthesia

* is receiving medication in a dose and/or at a time point known to

interfere with neuromuscular blocking agents (NMBAs), such as antibiotics, anticonvulsants and Mg2+

* already participated in a sugammadex trial
* participated in another clinical trial, not pre-approved, within prior 30 days
* pregnant females
* breast-feeding females

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

REFERENCES:
- [Result] Drobnik L, Sparr HJ, Thorn SE, Khuenl-Brady KS, Rietbergen H, Prins ME, Ullman J. A randomized simultaneous comparison of acceleromyography with a peripheral nerve stimulator for assessing reversal of rocuronium-induced neuromuscular blockade with sugammadex. Eur J Anaesthesiol. 2010 Oct;27(10):866-73. doi: 10.1097/EJA.0b013e32833b1b85. PMID 20523215

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugammadex 1.0 mg/kg, TOF-Watch® SX Dominant Arm: Participants received an intubating dose of 0.6 mg/kg rocuronium, followed by one or more maintenance doses of 0.15 mg/kg rocuronium, if necessary. Fifteen minutes after the last dose of rocuronium, 1.0 mg/kg sugammadex was administered by intravenous (IV) bolus dose based on actual body weight. The Train of Four (TOF)-Watch® SX was on the dominant forearm and the peripheral nerve stimulator (PNS) was on the non-dominant forearm.
- Sugammadex 1.0 mg/kg, TOF-Watch® SX Non-dominant Arm: Participants received an intubating dose of 0.6 mg/kg rocuronium, followed by one or more maintenance doses of 0.15 mg/kg rocuronium, if necessary. Fifteen minutes after the last dose of rocuronium, 1.0 mg/kg sugammadex was administered by intravenous (IV) bolus dose based on actual body weight. The TOF-Watch® SX was on the non-dominant forearm and the PNS was on the dominant forearm.
- Sugammadex 4.0 mg/kg, TOF-Watch® SX Dominant Arm: Participants received an intubating dose of 0.6 mg/kg rocuronium, followed by one or more maintenance doses of 0.15 mg/kg rocuronium, if necessary. Fifteen minutes after the last dose of rocuronium, 4.0 mg/kg sugammadex was administered by intravenous (IV) bolus dose based on actual body weight. The TOF-Watch® SX was on the dominant forearm and the PNS was on the non-dominant forearm.
- Sugammadex 4.0 mg/kg, TOF-Watch® SX Non-dominant Arm: Participants received an intubating dose of 0.6 mg/kg rocuronium, followed by one or more maintenance doses of 0.15 mg/kg rocuronium, if necessary. Fifteen minutes after the last dose of rocuronium, 4.0 mg/kg sugammadex was administered by intravenous (IV) bolus dose based on actual body weight. The TOF-Watch® SX was on the non-dominant forearm and the PNS was on the dominant forearm.
Period: Overall Study
Arm/Group | Sugammadex 1.0 mg/kg, TOF-Watch® SX Dominant Arm | Sugammadex 1.0 mg/kg, TOF-Watch® SX Non-dominant Arm | Sugammadex 4.0 mg/kg, TOF-Watch® SX Dominant Arm | Sugammadex 4.0 mg/kg, TOF-Watch® SX Non-dominant Arm
Started | 15 | 15 | 30 | 31
All-Subjects-Treated (AST) Group | 15 | 14 | 30 | 31
Completed | 15 | 13 | 30 | 31
Not Completed | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Not treated with sugammadex | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sugammadex 1.0 mg/kg: Participants received an intubating dose of 0.6 mg/kg rocuronium, followed by one or more maintenance doses of 0.15 mg/kg rocuronium, if necessary. Fifteen minutes after the last dose of rocuronium, 1.0 mg/kg sugammadex was administered by intravenous (IV) bolus dose based on actual body weight.
- Sugammadex 4.0 mg/kg: Participants received an intubating dose of 0.6 mg/kg rocuronium, followed by one or more maintenance doses of 0.15 mg/kg rocuronium, if necessary. Fifteen minutes after the last dose of rocuronium, 4.0 mg/kg sugammadex was administered by intravenous (IV) bolus dose based on actual body weight.
- Total: Total of all reporting groups
Arm/Group | Sugammadex 1.0 mg/kg | Sugammadex 4.0 mg/kg | Total
Number analyzed (Participants) | 29 | 61 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] — Randomization into dominant and non-dominant forearms was aimed at preventing bias; so differences between dominant and non-dominant forearms were not analyzed.
  years | 43 (11) | 42 (13) | 42 (12)
Sex: Female, Male [Count of Participants; unit: Participants] — Randomization into dominant and non-dominant forearms was aimed at preventing bias; so differences between dominant and non-dominant forearms were not analyzed.
  Participants
    Female | 16 | 40 | 56
    Male | 13 | 21 | 34

OUTCOME MEASURES:

1. Primary Outcome: Time From Start of Administration of 4.0 mg/kg Sugammadex to Recovery of the T4/T1 Ratio to 0.9 Measured by a TOF-Watch® SX
Description: Neuromuscular function was monitored by applying repetitive TOF electrical stimulations with the TOF-Watch® SX to the ulnar nerve of one forearm every 15 seconds & assessing twitch response at the adductor pollicis muscle with the TOF-Watch® SX. T1 and T4 are the magnitudes (heights) of the first and fourth twitches respectively after TOF nerve stimulation, where stimulation was continued until the T4/T1 ratio reached 0.9. A higher T4/T1 ratio indicates a lower degree of neuromuscular blockade, with a value of 1.0 representing full recovery. Only participants treated with 4.0 mg/kg sugammadex are presented, where the TOF-Watch® SX on the dominant forearm n =30, and on the non-dominant forearm n = 31. The 1.0 mg/kg sugammadex group was not evaluated for this outcome measure.
Time Frame: Up to 4 minutes after administering sugammadex
Population: The Intent-To-Treat (ITT) population: randomized, received 4.0 mg/kg sugammadex, and had at least one efficacy measurement. As dominant and non-dominant forearms were aimed at preventing bias, their differences were not analyzed. One participant who did not reach a T4/T1 ratio of 0.9 was not analyzed.The 1.0 mg/kg group was not evaluated.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex 4.0 mg/kg
Number analyzed (Participants) | 60
Minutes | 1.5 (0.7) [82 to 102]

2. Other Pre Specified Outcome: Time From Start of Administration of 1.0 mg/kg Sugammadex to Recovery of the T4/T1 Ratio to 0.9 Measured by a TOF-Watch® SX
Description: Neuromuscular function was monitored by applying repetitive TOF electrical stimulations with the TOF-Watch® SX to the ulnar nerve of one forearm every 15 seconds & assessing twitch response at the adductor pollicis muscle with the TOF-Watch® SX. T1 and T4 are the magnitudes (heights) of the first and fourth twitches respectively after TOF nerve stimulation, where stimulation was continued until the T4/T1 ratio reached 0.9. A higher T4/T1 ratio indicates a lower degree of neuromuscular blockade, with a value of 1.0 representing full recovery. Only participants treated with 1.0 mg/kg sugammadex are presented where the TOF-Watch® SX on the dominant forearm n =15, and on the non-dominant forearm n = 14. The 4.0 mg/kg sugammadex group was not evaluated for this outcome measure.
Time Frame: Up to 150 minutes after administering sugammadex
Population: The ITT population: randomized participants who received 1.0 mg/kg sugammadex, and had at least one efficacy measurement. As dominant and non-dominant forearms were aimed at preventing bias, their differences were not analyzed. One participant was not analyzed as the time of recovery was judged unreliable. The 4.0 mg/kg group was not evaluated.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex 1.0 mg/kg
Number analyzed (Participants) | 28
Minutes | 17.2 (28.6)

3. Other Pre Specified Outcome: Time From Start of Administration of 1.0 or 4.0 mg/kg Sugammadex to Reappearance of T4 Measured by a TOF-Watch® SX
Description: Neuromuscular function was monitored by applying repetitive TOF electrical stimulations with the TOF-Watch® SX to the ulnar nerve of one forearm every 15 seconds & assessing twitch response at the adductor pollicis muscle with the TOF-Watch® SX. T4 is the fourth twitch after TOF nerve stimulation. For participants treated with 1.0 mg/kg sugammadex the TOF-Watch® SX on the dominant forearm n =15, and on the non-dominant forearm n = 14. For participants treated with 4.0 mg/kg sugammadex the TOF-Watch® SX on the dominant forearm n =30, and on the non-dominant forearm n = 31.
Time Frame: Up to 7 minutes after administering sugammadex
Population: The ITT population consisting of all randomized participants who received 1.0 or 4.0 mg/kg sugammadex, and had at least one efficacy measurement. As dominant and non-dominant forearms were aimed at preventing bias, their differences were not analyzed.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex 1.0 mg/kg | Sugammadex 4.0 mg/kg
Number analyzed (Participants) | 29 | 61
Minutes | 2.1 (1.6) | 0.8 (0.2)

4. Other Pre Specified Outcome: Time From Start of Administration of 1.0 mg/kg Sugammadex to Reappearance of T4 Measured by a PNS
Description: Neuromuscular function was monitored by applying repetitive TOF stimulations manually to the ulnar nerve of one forearm every 15 seconds & the number of twitches collected manually at the adductor pollicis muscle with the PNS by a blinded PNS assessor. T4 is the fourth twitch after TOF nerve stimulation. Only participants treated with 1.0 mg/kg sugammadex are presented, where the PNS on the dominant forearm n =15, and on the non-dominant forearm n = 14. The 4.0 mg/kg sugammadex group was not evaluated for this outcome measure.
Time Frame: Up to 5 minutes after administering sugammadex
Population: The ITT population consisting of all randomized participants who received 1.0 mg/kg sugammadex, and had at least one efficacy measurement. As dominant and non-dominant forearms were aimed at preventing bias, their differences were not analyzed. Participants treated with 4.0 mg/kg were not evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex 1.0 mg/kg
Number analyzed (Participants) | 29
Minutes | 1.7 (1.1)

5. Other Pre Specified Outcome: Time From Start of Administration of 1.0 or 4.0 mg/kg Sugammadex to Recovery of the T4/T1 Ratio to 0.8 Measured by a TOF-Watch® SX
Description: Neuromuscular function was monitored by applying repetitive TOF electrical stimulations with the TOF-Watch® SX to the ulnar nerve of one forearm every 15 seconds & assessing twitch response at the adductor pollicis muscle with the TOF-Watch® SX. T1 and T4 are the magnitudes (heights) of the first and fourth twitches respectively after TOF nerve stimulation, where stimulation was continued until the T4/T1 ratio reached 0.8. A higher T4/T1 ratio indicates a lower degree of neuromuscular blockade, with a value of 1.0 representing full recovery. For participants treated with 1.0 mg/kg sugammadex the TOF-Watch® SX on the dominant forearm n =15, and on the non-dominant forearm n = 14. For participants treated with 4.0 mg/kg sugammadex the TOF-Watch® SX on the dominant forearm n =30, and on the non-dominant forearm n = 31.
Time Frame: Up to 42 minutes after administering sugammadex
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex 1.0 mg/kg | Sugammadex 4.0 mg/kg
Number analyzed (Participants) | 29 | 61
Minutes | 9.9 (11.4) | 1.3 (1.4)

6. Other Pre Specified Outcome: Time From Start of Administration of 1.0 or 4.0 mg/kg Sugammadex to Recovery of the T4/T1 Ratio to 0.7 Measured by a TOF-Watch® SX
Description: Neuromuscular function was monitored by applying repetitive TOF electrical stimulations with the TOF-Watch® SX to the ulnar nerve of one forearm every 15 seconds & assessing twitch response at the adductor pollicis muscle with the TOF-Watch® SX. T1 and T4 are the magnitudes (heights) of the first and fourth twitches respectively after TOF nerve stimulation, where stimulation was continued until the T4/T1 ratio reached 0.7. A higher T4/T1 ratio indicates a lower degree of neuromuscular blockade, with a value of 1.0 representing full recovery. For participants treated with 1.0 mg/kg sugammadex the TOF-Watch® SX on the dominant forearm n =15, and on the non-dominant forearm n = 14. For participants treated with 4.0 mg/kg sugammadex the TOF-Watch® SX on the dominant forearm n =30, and on the non-dominant forearm n = 31.
Time Frame: Up to 42 minutes after administering sugammadex
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex 1.0 mg/kg | Sugammadex 4.0 mg/kg
Number analyzed (Participants) | 29 | 61
Minutes | 7.6 (10.2) | 1.1 (0.9)

7. Primary Outcome: Time From Start of Administration of 4.0 mg/kg Sugammadex to Reappearance of T4 Measured by a Peripheral Nerve Stimulator (PNS)
Description: Neuromuscular function was monitored with a PNS by applying repetitive TOF stimulation to the ulnar nerve of one forearm every 15 seconds and assessing the number of twitches at the adductor pollicis muscle by a blinded PNS assessor. T4 is the fourth twitch after TOF nerve stimulation. Only participants treated with 4.0 mg/kg sugammadex are presented, where the PNS on the dominant forearm n =31, and on the non-dominant forearm n = 30. The 1.0 mg/kg sugammadex group was not evaluated for this outcome measure.
Time Frame: up to 2 minutes after administering sugammadex
Population: The ITT population consisting of all randomized participants who received 4.0 mg/kg sugammadex, and had at least one efficacy measurement. As dominant and non-dominant forearms were aimed at preventing bias, their differences were not analyzed. Participants treated with 1.0 mg/kg were not evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex 4.0 mg/kg
Number analyzed (Participants) | 61
Minutes | 0.8 (0.3) [42 to 50]

8. Primary Outcome: Difference in Time Between Recovery of T4/T1 Ratio to 0.9 as Measured by TOF Watch® SX, and Reappearance of T4 as Measured by PNS, Within Participants, After Administration of 4.0 mg/kg Sugammadex
Description: The difference between the recovery of T4/T1 ratio to 0.9 and reappearance of T4 within participants was assessed from an ANOVA method. Only participants treated with 4.0 mg/kg sugammadex are presented, where the TOF-Watch® SX on the dominant forearm n =30, and on the non-dominant forearm n = 31; and the PNS on the dominant forearm n =31, and on the non-dominant forearm n = 30. The 1.0 mg/kg sugammadex group was not evaluated for this outcome measure.
Time Frame: Up to 3 minutes after administering sugammadex
Population: The ITT population: all randomized participants who received 4.0 mg/kg sugammadex, and had at least one efficacy measurement. As dominant and non-dominant forearms were aimed at preventing bias; their differences were not analyzed. One participant who did not reach a T4/T1 ratio of 0.9 was not analyzed. The 1.0 mg/kg group was not evaluated.
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Sugammadex 4.0 mg/kg
Number analyzed (Participants) | 60
Minutes | 0.8 (0.6) [0.6 to 0.9]

ADVERSE EVENTS:
Time Frame: From screening period up to and including seventh post-operative day
Description: All Patients Treated. One participant from the 1.0 mg/kg sugammadex group was not treated, and discontinued from the study.
Arm/Group | Sugammadex 1.0 mg/kg | Sugammadex 4.0 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/29 | 3/61
Other Adverse Events (participants affected / at risk) | 24/29 | 53/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex 1.0 mg/kg (N=29) | Sugammadex 4.0 mg/kg (N=61)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Perforation bile duct (Hepatobiliary disorders) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bladder disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex 1.0 mg/kg (N=29) | Sugammadex 4.0 mg/kg (N=61)
Nausea (Gastrointestinal disorders) | 8 (8) | 19 (19)
Vomiting (Gastrointestinal disorders) | 6 (6) | 9 (10)
Incision site pain (Injury, poisoning and procedural complications) | 8 (9) | 17 (18)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Procedural hypertension (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Procedural hypotension (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Procedural pain (Injury, poisoning and procedural complications) | 12 (14) | 31 (35)
Underdose (Injury, poisoning and procedural complications) | 7 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any scientific paper, presentation, or other communication concerning the clinical trial will first be submitted at least six weeks ahead of publication or presentation, for written consent. The Sponsor shall have the right to make its consent conditional upon proper representation of the interpretation and discussion of the data.